CLINICAL TRIAL: NCT06759363
Title: Exploring the Potential of Oral Butyrate Supplementation in Metabolic Dysfunction-Assosciated Steatotic Liver Disease Patients
Brief Title: MASLD Butyrate Supplementation Treatment Efficacy Review
Acronym: MASTER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Medical Center Zvezdara (Other)
Responsible Party: Principal Investigator, Miloš Mitrović, MD, Miloš Mitrović- digestive disease specialist at Gastroenterology and Hepatology Unit of Internal Medicine Clinic of University Medical center, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.11.24.
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-01

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Butyrate supplementation; MASLD; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Butyric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Butyrate Arm (Active Comparator): 1000 mg/day Sodium butyrate in combination with a Mediterranean diet during 12 weeks
  Interventions: Drug: Sodium-Butyrate
- Calcium Butyrate Arm (Active Comparator): 1000 mg/day calcium butyrate in combination with a Mediterranean diet during 12 weeks
  Interventions: Drug: Calcium Butyrate

INTERVENTIONS:
Drug: Sodium-Butyrate — 1000 mg/day of sodium-butyrate
  Other Names: Colosal
  Arms: Sodium Butyrate Arm
Drug: Calcium Butyrate — 1000 mg/day of calcium-butyrate
  Other Names: Dibuzin
  Arms: Calcium Butyrate Arm

SUMMARY:
1. Study Design This is an interventional study designed to evaluate the efficacy of oral butyrate supplementation in patients diagnosed with metabolic dysfunction-associated steatotic liver disease (MASLD).
2. Introduction MASLD is becoming an increasingly significant global public health issue, though the underlying mechanisms of this disorder are not fully understood. Emerging research highlights the crucial role of the gut microbiota, particularly through the production of short-chain fatty acids such as butyrate, in regulating metabolic processes related to MASLD. Animal studies have shown that butyrate has beneficial effects on liver function, but large-scale human studies exploring this potential are lacking. Butyrates have long been used in the treatment of irritable bowel syndrome without significant adverse effects.
3. Study Objectives

   Primary Objective:

   To assess the impact of oral butyrate supplementation on liver steatosis in patients with MASLD, measured by changes in the attenuation coefficient (ATT) using point shear wave elastography (pSWE).

   Secondary Objectives:
   * Evaluate changes in alanine aminotransferase (ALT) levels.
   * Assess the impact on inflammatory markers (high-sensitivity C-reactive protein [hsCRP], tumor necrosis factor-alpha [TNF-α], interleukin-1, interleukin-6, and cytokeratin-18).
   * Measure changes in lipid profile and stool short-chain fatty acids (SCFA).
   * Evaluate microRNA expression (miR-192, miR-885, miR-122).
4. Methods/Study Design 4.1 Study Population and Inclusion Criteria

   Inclusion Criteria:
   * Patients aged 18-70 years with confirmed MASLD based on:

     * ATT > 0.63 dB/cm/MHz measured by pSWE.
     * ALT level > 40 IU/L.
   * Patients capable of providing informed consent.

   Exclusion Criteria:
   * History of other liver diseases (e.g., viral hepatitis, alcoholic liver disease).
   * Current use of medications known to affect liver function (e.g., statins, corticosteroids).
   * Pregnant and breastfeeding women. 4.2 Sample Size and Power Calculation The study will include 200 patients with MASLD, randomly assigned in a 1:1 ratio to receive either calcium butyrate or sodium butyrate. A sample size of 200 patients was determined to ensure sufficient power to detect significant differences in primary and secondary outcomes with an alpha value of 0.05 and 80% power.

   4.3 Randomization and Blinding Participants will be randomly assigned to two groups using computer-generated randomization. The study will be single-blind, meaning that patients will not know which type of butyrate they receive.

   4.4 Interventions
   * Group 1 (Calcium Butyrate): 1000 mg/day calcium butyrate.
   * Group 2 (Sodium Butyrate): 1000 mg/day sodium butyrate.
   * Both groups will follow a Mediterranean diet (20-30 kcal/kg body weight; 35-40% fats, 20% protein, 40-45% carbohydrates).
   * Treatment will last for 12 weeks. 4.5 Outcome Measures

   Primary Outcome:

   • Change in liver steatosis measured by ATT after 12 weeks compared to baseline.

   Secondary Outcomes:
   * Changes in ALT, inflammatory markers (hsCRP, TNF-α, IL-1, IL-6, cytokeratin-18), lipid profile, and stool SCFA levels.
   * Changes in microRNA expression (miR-192, miR-885, miR-122).
5. Data Collection and Analysis 5.1 Data Collection At baseline and after 12 weeks, the following assessments will be conducted:

   * Liver steatosis measured by pSWE.
   * Blood samples for ALT, inflammatory markers, and lipid profile.
   * Stool samples for SCFA analysis.
   * MicroRNA panel analysis (miR-192, miR-885, miR-122). 5.2 Statistical Analysis Data will be analyzed using SPSS software (v. XX). Baseline and 12-week data will be compared using paired t-tests or Wilcoxon tests. ANOVA will be used to assess differences between groups. Statistical significance will be set at p < 0.05.
6. Ethics and Dissemination 6.1 Ethical Considerations The study protocol has been submitted for review by the Ethics Committee of the Clinical Center of Serbia, Belgrade. Written consent will be obtained from all participants.

6.2 Data Management All patient data will be anonymized, securely stored, and managed following local data protection regulations.

6.3 Dissemination The study results will be published in peer-reviewed scientific journals and presented at international conferences. No commercial application of the results is planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years with confirmed MASLD based on:

ATT > 0.63 dB/cm/MHz measured by pSWE.

ALT level > 40 IU/L.

* Patients capable of providing informed consent.

Exclusion Criteria:

* History of other liver diseases (e.g., viral hepatitis, alcoholic liver disease).
* Current use of medications known to affect liver function (e.g., statins, corticosteroids).
* Pregnant and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in liver steatosis measured by ATT after 12 weeks compared to baseline | 12 weeks
  Liver steatosis is going to be assessed by the attenuation coefficient (ATT) on ultrasound B mode at two points- before the treatment and after the last drug dose, and define the absolute and relative change of this parameter.

SECONDARY OUTCOMES:
Changes in ALT and serum inflammatory markers (hsCRP, TNF-α, IL-1, IL-6, cytokeratin-18), lipid profile | 12 weeks
  Absolute and relative changes in ALT, inflammatory markers (hsCRP, TNF-α, IL-1, IL-6, cytokeratin-18), lipid profile between baseline and endpoint values will be assessed
Changes in stool SCFA levels. | 12 weeks
  Absolute and relative changes in stool SCFA levels between baseline and endopint will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Miloš V Mitrović, MD PhD, Principal Investigator — University Medical Center Zvezdara
Locations (1):
- University Medical Center Zvezdara, Belgrade, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Will make figshare.com repository of data, excluding patients personal data, and share it within publication

REFERENCES:
- [Background] Fogacci F, Giovannini M, Di Micoli V, Grandi E, Borghi C, Cicero AFG. Effect of Supplementation of a Butyrate-Based Formula in Individuals with Liver Steatosis and Metabolic Syndrome: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Nutrients. 2024 Jul 28;16(15):2454. doi: 10.3390/nu16152454. PMID 39125336